CLINICAL TRIAL: NCT00301028
Title: Phase II Trial of Induction Therapy With Cetuximab (C225) and Carboplatin/Paclitaxel Chemotherapy in Previously Untreated Patients With Advanced (Stage IV) Head & Neck Squamous Cell Carcinoma
Brief Title: Cetuximab, Carboplatin, and Paclitaxel Followed by Radiation Therapy, With or Without Cisplatin, in Treating Patients With Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0919; P50CA097007 (NIH); P30CA016672 (NIH); MDA-2003-0919 (Other: UT MD Anderson Cancer Center); BMS-CA225054; CDR0000441273 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Results first posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-02

CONDITIONS: Head and Neck Cancer
Keywords: stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the lip and oral cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab + Carboplatin/Paclitaxel (Experimental): Cetuximab beginning weekly dose 400 mg/m^2 intravenous (IV), and 250 mg/m^2 weeks 2-6; Weekly Carboplatin area under the curve (AUC) 2 and Paclitaxel 135 mg/m^2 for 6 courses.
  Interventions: Biological: Cetuximab; Drug: Carboplatin; Drug: Paclitaxel; Procedure: Conventional Surgery; Radiation: Radiation Therapy

INTERVENTIONS:
Biological: Cetuximab — Beginning weekly dose 400 mg/m^2 IV over 1-2 hours, and 250 mg/m^2 weeks 2-6.
  Other Names: C225; Erbitux; IMC-C225
Drug: Carboplatin — AUC 2 weekly for 6 courses.
  Other Names: Paraplatin
Drug: Paclitaxel — 135 mg/m^2 weekly for 6 courses.
  Other Names: Taxol
Procedure: Conventional Surgery — Following induction in second part of study.
Radiation: Radiation Therapy — Following induction in second part of study.
  Other Names: Radiotherapy; RT; XRT

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as carboplatin, paclitaxel, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells. Giving cetuximab together with combination chemotherapy and radiation therapy, with or without cisplatin, may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab together with carboplatin and paclitaxel followed by radiation therapy, with or without cisplatin, works in treating patients with metastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the increase in clinical/radiographic complete response rate in patients with previously untreated metastatic squamous cell carcinoma of the head and neck treated with induction therapy comprising cetuximab, carboplatin, and paclitaxel.
* Determine the toxic effects of this regimen in these patients.

Secondary

* Determine the pattern of tumor recurrence in patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.
* Determine the duration of response, time to progression, and survival of patients treated with this regimen.
* Correlate effects of this regimen with biomarkers of response and predictors of long-term outcome in these patients.

OUTLINE: This is a nonrandomized, open-label study.

Patients receive induction therapy comprising cetuximab IV over 1-2 hours, paclitaxel IV over 1 hour, and carboplatin IV over 1 hour on day 1. Treatment repeats weekly for up to 6 courses in the absence of disease progression or unacceptable toxicity. Beginning 2-3 weeks later, patients undergo radiotherapy or chemoradiotherapy. Patients with T0, 1, 2 disease undergo radiotherapy 5 days a week for 6 weeks. Patients with T3, 4 disease or unresectable nodal disease undergo radiotherapy 5 days a week for 6 weeks and receive concurrent cisplatin IV over 1-2 hours on days 1 and 22. Some patients may undergo primary surgical resection before or instead of radiotherapy or chemoradiotherapy.

Quality of life is assessed at baseline and at 6, 12, and 24 months after completion of radiotherapy or surgery.

After study completion, patients are followed every 3 months for 2 years, every 4 months for 1 year, and every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological proof (from the primary lesion and/or lymph nodes) of squamous cell carcinoma of the oral cavity, oropharynx, nasopharynx, hypopharynx, or larynx.
2. Patients should have stage IV disease, stage T0-4 N2b/2c/3 M0 (for nasopharynx patients, stage N1 disease is eligible). Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) is required.
3. Patients with stage Tx primary disease are eligible if there is N2b/3 adenopathy.
4. Karnofsky performance status of >/= 80 or Eastern Cooperative Oncology Group (ECOG) point scale 0-1
5. Age > 16 years
6. Patients should have adequate bone marrow function defined as an absolute peripheral granulocyte count (AGC) of > 1500 cells/mm3 and platelet count of > 100,000 cells/mm3; adequate hepatic function with bilirubin </= Upper Limit of Normal (ULN), aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) may be up to 2.5 times the upper limit of normal if alkaline phosphatase is normal. Alkaline phosphatase may be up to 4* ULN if SGPT and SGOT are normal. Patients who have both SGPT and SGOT > 1.5 ULN and alkaline phosphatase > 2.5 * ULN are not eligible. Normal PT/PTT and normal serum calcium (without intervention) are required.
7. Creatinine clearance > 40 ml/min determined by 24 hour collection or nomogram: CrCl male = (140 - age) times (weight in kg)/serum Cr times 72 CrCl female = 0.85 times (CrCl male)
8. Patients should have no serious acute or chronic co-morbid condition, or acute infection.
9. Patients must sign a study-specific informed consent form.

Exclusion Criteria:

1. Histology other than squamous cell carcinoma.
2. Evidence of distant metastases (below the clavicle) by clinical or radiographic means.
3. Karnofsky performance status < 80 or ECOG>1
4. Prior chemotherapy, within the previous 3 years.
5. Prior radiotherapy to the head and neck.
6. Prior cetuximab therapy, prior therapy with any other drug that targets the EGFR pathway, or prior therapy with a murine or chimeric monoclonal antibody.
7. Initial surgical resection rendering the patient clinically and radiologically disease free.
8. Simultaneous primary invasive cancers.
9. Patients with another malignancy (excluding non melanoma skin cancers, and cancers treated > 3 years prior for which patient remains continuously disease free).
10. Women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the study. Subjects who are men must also agree to use effective contraception. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin (HCG)) within 72 hours prior to the start of study medication.
11. WOCBP using a prohibited contraceptive method.
12. Women who are pregnant or breastfeeding.
13. Women with a positive pregnancy test on enrollment or prior to study drug administration.
14. Refusal to sign the informed consent.
15. Pre-existing peripheral neuropathy Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or worse.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merrill S. Kies, MD, Study Chair — M.D. Anderson Cancer Center; Vassiliki A. Papadimitrakopoulou, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center at University of Texas, Houston, Texas, United States

REFERENCES:
- [Result] Kies MS, Holsinger FC, Lee JJ, William WN Jr, Glisson BS, Lin HY, Lewin JS, Ginsberg LE, Gillaspy KA, Massarelli E, Byers L, Lippman SM, Hong WK, El-Naggar AK, Garden AS, Papadimitrakopoulou V. Induction chemotherapy and cetuximab for locally advanced squamous cell carcinoma of the head and neck: results from a phase II prospective trial. J Clin Oncol. 2010 Jan 1;28(1):8-14. doi: 10.1200/JCO.2009.23.0425. Epub 2009 Nov 16. PMID 19917840
- [Derived] Psyrri A, Rampias T, Vermorken JB. The current and future impact of human papillomavirus on treatment of squamous cell carcinoma of the head and neck. Ann Oncol. 2014 Nov;25(11):2101-2115. doi: 10.1093/annonc/mdu265. Epub 2014 Jul 23. PMID 25057165
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 31, 2005 to September 16, 2011
Pre-assignment Details: Of the forty-eight (48) participants registered, forty-seven (47) were eligible to participate in this trial
Period: Overall Study
Arm/Group | Cetuximab + Carboplatin/Paclitaxel
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cetuximab + Carboplatin/Paclitaxel: Cetuximab beginning weekly dose 400 mg/m^2 intravenous (IV), and 250 mg/m^2 weeks 2-6; Weekly Carboplatin AUC 2 and Paclitaxel 135 mg/m^2 for 6 courses.
Arm/Group | Cetuximab + Carboplatin/Paclitaxel
Number analyzed (Participants) | 47
Age Continuous [Median (Full Range); unit: years] | 53 [21 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response
Description: Number of participants with a complete response. Complete Response (CR): Disappearance of clinical and radiological evidence of tumor.
Time Frame: Study period of 3 Years
Measure: Number; unit: participants
Arm/Group | Cetuximab + Carboplatin/Paclitaxel
Number analyzed (Participants) | 47
participants | 39

ADVERSE EVENTS:
Time Frame: 6 years
Arm/Group | Cetuximab + Carboplatin/Paclitaxel
Serious Adverse Events (participants affected / at risk) | 37/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab + Carboplatin/Paclitaxel (N=47)
Anorexia (Psychiatric disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 11
Mucositis (Gastrointestinal disorders) | 37
Fatigue (General disorders) | 3
Rash/folliculitis (Skin and subcutaneous tissue disorders) | 21
Sensory neuropathy (Nervous system disorders) | 1
Allergic reaction (Investigations) | 2
Dry mouth (General disorders) | 2
Taste alteration (General disorders) | 2
Dehydration (Gastrointestinal disorders) | 3
Nausea/vomiting (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab + Carboplatin/Paclitaxel (N=47)
Arthralgia/myalgia (General disorders) | 6
Anorexia (Psychiatric disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 19
Nausea/vomiting (Gastrointestinal disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash/folliculitis (Skin and subcutaneous tissue disorders) | 6
Sensory neuropathy (Nervous system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 11
Anemia (Blood and lymphatic system disorders) | 4
Dry mouth (General disorders) | 14
Taste alteration (General disorders) | 15
Mucositis (Gastrointestinal disorders) | 7
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6
Tinnitus (Ear and labyrinth disorders) | 3
Sensory neuropathy (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No